CLINICAL TRIAL: NCT01265823
Title: Immediate Response With Adalimumab and Its Impact on Quality of Life and Other Comorbidity Factors in Patients With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W11-050
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-02

CONDITIONS: Psoriasis
Keywords: Humira; Adalimumab; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab (Experimental)
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Adalimumab was administered as follows: 80 mg at baseline, followed by 40 mg every other week (eow; starting at Week 1 until Week 15). The study drug was self-administered via subcutaneous (sc) injection.
  Other Names: ABT-D2E7; Humira

SUMMARY:
W11-050 is a Mexican open label multicenter study that has been designed to further assess the safety and efficacy of adalimumab in the treatment of patients with active plaque psoriasis who have failed prior conventional systemic psoriasis treatment or who are candidates for systemic therapy.

DETAILED DESCRIPTION:
Up to 150 subjects having a diagnosis of active plaque psoriasis and fulfilling the study eligibility criteria were enrolled in Mexico. Adalimumab was administered as follows: 80 mg at baseline, followed by 40 mg every other week (eow; starting at week 1 until week 15). The study drug was self administered via subcutaneous (sc) injection. Safety and efficacy measures were performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent prior to any study related procedures and to comply with the requirements of the study protocol
2. Male and female subjects between 18 and 75 years old
3. Diagnosis of moderate to severe types I and II plaque psoriasis (Type I : symptoms onset before 40 years old; Type II: symptoms onset after 40 years old), with at least 6 months of duration
4. Documented moderate to severe plaque psoriasis based on Psoriasis Area and Severity Index (PASI) score >10
5. Subjects naïve to adalimumab therapy
6. Subject must be evaluated for active and latent tuberculosis (TB) infection by using a Purified Protein Derivative (PPD) skin test, chest x-ray (posterior to anterior (PA) and lateral views) and a detailed review of the subject's medical history. This screening must be negative
7. A negative pregnancy test (serum human chorionic gonadotrophin) for women of childbearing potential prior to start of study treatment. (Non-childbearing potential is defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy])
8. Able and willing to self-administer subcutaneous injections or have available a suitable person to administer subcutaneous injections
9. Subject is judged to be in generally good health as determined by the investigator

Exclusion Criteria:

1. Prior treatment with any investigational agent within 30 days, or five half-lives of the product, which ever is longer. Subject has been treated with any investigational drug of chemical or biologic nature within a minimum of 30 days or five half lives (whichever is longer) of the drug prior to study entry (Baseline Visit)
2. Subject has other active skin diseases or skin infections (bacterial, fungal, or viral) that may interfere with the evaluation of psoriasis or compromise the subject's safety
3. Subject has a history of dysplasia, malignancy (including lymphoma and leukemia), or lymphoproliferative disease other than: a. Successfully and completely treated non-metastatic squamous or basal cell carcinoma of the skin with no recurrence within the last five years. b. Localized carcinoma in situ of the cervix or cervical dysplasia, with no recurrence within the last five years
4. Persistent or recurrent infections or severe infections requiring hospitalization or treatment with intravenous (IV) antibiotics, IV antivirals, or IV antifungals within 30 days, or oral antibiotics, oral antivirals or oral antifungals within 14 days prior to Baseline Visit
5. Other medical conditions: uncontrolled diabetes, unstable ischemic heart disease, congestive heart failure New York Heart Association (NYHA) III-IV, recent stroke (within three months), chronic leg ulcer and any other condition (e.g., indwelling urinary catheter) which, in the opinion of the investigator, may place the subject at risk
6. Previous diagnosis or signs highly indicative of central nervous system demyelinating diseases (e.g., optic neuritis, ataxia, apraxia)
7. History of listeriosis, histoplasmosis, chronic or active Hepatitis B infection, human immunodeficiency virus (HIV) infection, immunodeficiency syndrome, chronic recurring infections or active TB
8. Female subjects who are pregnant or breast-feeding
9. History of clinically significant drug or alcohol abuse in the last year
10. Subject started receiving a new topical therapy within the last four weeks prior to the Baseline visit for areas other than the palms, soles of feet, axilla and groin
11. Subject started being treated with ultraviolet B (UVB) phototherapy, within the last four weeks prior to the Baseline visit
12. Subject was treated with psoralen ultraviolet A (PUVA) phototherapy within the last four weeks prior to the Baseline visit
13. Subject has been initiated on a new systemic agent within the last four weeks prior to the Baseline visit
14. Patients with history of atopy
15. Patients with any other autoimmune disease such as systemic lupus erythematosus (SLE) , Sdx Sjögren, vasculitis etc
16. Known hypersensitivity to the excipients of adalimumab as stated in the label
17. Female subjects who are pregnant or breast-feeding or considering becoming pregnant during the study
18. Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study
19. Subject with any prior exposure to Tysabri (natalizumab), or Orencia (abatacept)
20. Subjects with positive immunologic test for hepatitis A, B or C (Positive test of any of the following: hepatitis A viral antibody immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab)
21. Subjects with a positive immunologic test for HIV determined by enzyme-linked immunosorbent assay (ELISA) method

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose-Luis Canadas, Medical Director, MD, Study Director — AbbVie
Locations (8):
- Mexico (8):
  - Site Reference ID/Investigator# 50942, Circuito Comercial Satelite
  - Site Reference ID/Investigator# 40964, Iztapalapa
  - Site Reference ID/Investigator# 50943, Mexico City
  - Site Reference ID/Investigator# 40965, Monterrey
  - Site Reference ID/Investigator# 40962, Monterrey
  - Site Reference ID/Investigator# 40662, Toluca
  - Site Reference ID/Investigator# 41062, Toluca
  - Site Reference ID/Investigator# 40963, Zapopan

REFERENCES:
- See also: Related info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 187 participants were screened and 37 were considered screening failures.
Period: Overall Study
Arm/Group | Adalimumab
Started | 150
Completed | 143
Not Completed | 7
Not completed — Unsatisfactory Response Efficacy | 1
Not completed — Failure to Return | 4
Not completed — Protocol Violation | 1
Not completed — Participant Request | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 150
Age Continuous [Mean (Standard Deviation); unit: years] | 44.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 113
Region of Enrollment [Number; unit: participants]
  Mexico | 150

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Psoriasis Area and Severity Index (PASI)-75 Response at Week 4
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 4. The improvement in PASI score was used as a measure of efficacy.
Time Frame: Week 4
Population: Intention-to-treat (ITT) population. Participants with missing scores were considered nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 150
percentage of participants | 31

2. Primary Outcome: Percentage of Participants With Psoriasis Area and Severity Index (PASI)-75 Response at Week 16
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI-75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 16. The improvement in PASI score was used as a measure of efficacy.
Time Frame: Week 16
Population: Intention-to-treat (ITT) population. Participants with missing scores were considered nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 150
percentage of participants | 85

3. Primary Outcome: Percentage of Participants With a Dermatology Life Quality Index (DLQI) Score < 6 at Week 4
Description: Dermatology Life Quality Index (DLQI) score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot, a little, or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired. A score <6 indicates that psoriasis has small or no effect at all on participant's life.
Time Frame: Week 4
Population: Intention-to-treat (ITT) population. Participants with missing scores were considered nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 150
percentage of participants | 65

4. Primary Outcome: Percentage of Participants With a Dermatology Life Quality Index (DLQI) Score < 6 at Week 16
Description: as for outcome 3
Time Frame: Week 16
Population: Intention-to-treat (ITT) population. Participants with missing scores were considered nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 150
percentage of participants | 86

5. Secondary Outcome: Mean Score of Dermatology Life Quality Index (DLQI) at Baseline and Week 4
Description: Dermatology Life Quality Index (DLQI) score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot, a little, or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired.
Time Frame: Baseline, Week 4
Population: Participants with evaluable data at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 148
units on a scale
  Score at Baseline | 11.7 (6.3)
  Score at Week 4 | 5.2 (6.4)

6. Secondary Outcome: Mean Score of Dermatology Life Quality Index (DLQI) at Baseline and Week 16
Description: as for outcome 5
Time Frame: Baseline, Week 16
Population: Participants with evaluable data at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 143
units on a scale
  Score at Baseline | 11.7 (6.3)
  Score at Week 16 | 1.8 (2.0)

7. Secondary Outcome: Dermatology Life Quality Index (DLQI) Categories at Week 4
Description: Dermatology Life Quality Index (DLQI) score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot, a little, or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired. The following scoring categories present the effect on participant's life: 0-1 no effect at all; 2-5 small effect; 6-10 moderate effect; 11-20 very large effect; 21-30 extremely large effect.
Time Frame: Week 4
Population: ITT population. Participants with missing scores were considered nonresponders.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 150
participants
  No Effect | 42
  Small Effect | 52
  Moderate Effect | 32
  Very Large Effect | 18
  Extremely Large Effect | 3
  Missing | 3

8. Secondary Outcome: Dermatology Life Quality Index (DLQI) Categories at Week 16
Description: as for outcome 7
Time Frame: Week 16
Population: ITT population. Participants with missing scores were considered nonresponders.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 150
participants
  No Effect | 105
  Small Effect | 18
  Moderate Effect | 15
  Very Large Effect | 6
  Extremely Large Effect | 0
  Missing | 6

9. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI)-50, 90, 100 Responses at Week 4
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI-50, 90, and 100 responses are the percentage of participants who achieved at least a 50%, 90%, or 100% reduction (improvement) from baseline in PASI score at Week 4. 100% reduction was considered complete clearance of psoriasis.
Time Frame: Week 4
Population: ITT population. Participants with missing scores were considered nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 150
percentage of participants
  PASI-50 | 58.6
  PASI-90 | 10.6
  PASI-100 | 2.0

10. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI)-50, 90, 100 Responses at Week 16
Description: as for outcome 9
Time Frame: Week 16
Population: ITT population. Participants with missing scores were considered nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 150
percentage of participants
  PASI-50 | 92.6
  PASI-90 | 73.3
  PASI-100 | 49.3

11. Secondary Outcome: Physician's Global Assessment (PGA) at Week 4
Description: The PGA is a 7-point scale used to measure the severity of disease at the time of the physician's evaluation of the participant. Categories are as follows: Severe = very marked plaque elevation, scaling, and/or erythema; Moderate to severe = marked plaque elevation, scaling, and/or erythema; Moderate = moderate plaque elevation, scaling, and/or erythema; Mild to moderate = intermediate between moderate and mild; Mild = slight plaque elevation, scaling, and/or erythema; Almost clear = intermediate between mild and clear; Clear = no signs of psoriasis (post-inflammatory hypopigmentation or hyperpigmentation could be present).
Time Frame: Week 4
Population: ITT population. Participants with missing scores were considered nonresponders.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 150
participants
  Severe | 3
  Moderate to Severe | 12
  Moderate | 44
  Mild to Moderate | 37
  Mild | 36
  Almost Clear | 11
  Clear | 3
  Missing | 4

12. Secondary Outcome: Physician's Global Assessment (PGA) at Week 16
Description: The PGA is a 7-point scale used to measure the severity of disease at the time of the physician's evaluation of the participant. Categories are as follows: Severe = very marked plaque elevation, scaling, and/or erythema; Moderate to severe = marked plaque elevation, scaling, and/or erythema; Moderate = moderate plaque elevation, scaling, and/or erythema; Mild to moderate = intermediate between moderate and mild; Mild = slight plaque elevation, scaling, and/or erythema; Almost clear = intermediate between mild and clear; Clear = no signs of psoriasis (post-inflammatory hypopigmentation or hyperpigmentation could be present). The number of participants who achieve a PGA of 'clear' or 'almost clear' at Week 16 was a secondary outcome measure in this study.
Time Frame: Week 16
Population: ITT population. Participants with missing scores were considered nonresponders.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 150
participants
  Severe | 1
  Moderate to Severe | 1
  Moderate | 9
  Mild to Moderate | 8
  Mild | 9
  Almost Clear | 44
  Clear | 71
  Missing | 7

13. Secondary Outcome: Mean Lipid Profile, Triglycerides, and C-Reactive Protein (CRP) at Baseline and Week 16
Description: Normal values: C-reactive protein (CRP) 0-0.79 mg/dL; cholesterol 30-199 mg/dL; high density lipoprotein (HDL) 40-100 mg/dL; very low density lipoprotein (VLDL) 0-34 mg/dL; low density lipoprotein (LDL) 20-99 mg/dL; triglycerides 50-149 mg/dL.
Time Frame: Baseline, Week 16
Population: Participants with available data at given time points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adalimumab
Number analyzed (Participants) | 144
mg/dL
  C-reactive Protein at Baseline | 0.6 (0.9)
  C-reactive Protein at Week 16 | 0.5 (1.6)
  Cholesterol at Baseline | 190.7 (38.8)
  Cholesterol at Week 16 | 185.3 (33.8)
  High Density Lipoprotein (HDL) at Baseline | 41.6 (9.7)
  High Density Lipoprotein (HDL) at Week 16 | 42.6 (10.8)
  Very Low Density Lipoprotein (VLDL) at Baseline | 37.7 (26.3)
  Very Low Density Lipoprotein (VLDL) at Week 16 | 37.8 (20.9)
  Low Density Lipoprotein (LDL) at Baseline | 120.8 (28.7)
  Low Density Lipoprotein (LDL) at Week 16 | 120.3 (29.9)
  Triglycerides at Baseline | 185.3 (123.1)
  Triglycerides at Week 16 | 189.1 (104.3)

14. Secondary Outcome: Mean Homocysteine Levels at Baseline and Week 16
Description: Normal values for homocysteine were 5-13.9 µmol/L.
Time Frame: Baseline, Week 16
Population: Participants with available data at given time points.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 143
µmol/L
  Baseline | 11.6 (4.3)
  Week 16 | 10.9 (4.0)

15. Secondary Outcome: Percentage of Obese vs. Non-obese (Per Body Mass Index [BMI]) Participants Achieving a Psoriasis Area and Severity Index (PASI)-75 Response and a Total Dermatology Life Quality Index (DLQI) Score of <6 at Week 16
Description: The Body Mass Index (BMI) was used to determine the groups of participants who were overweight and who were considered obese. A BMI of 18.5 to 25 was considered normal range, 25 to 30 as overweight and 30 and above as obesity, in both men and women. Response to treatment in participants with obesity (based on Body Mass Index) versus those without obesity was assessed via PASI-75 response (see Outcome Measure 1 for details) and DLQI score of <6 (see Outcome Measure 3 for details).
Time Frame: Week 16
Population: ITT Population
Measure: Number; unit: percentage of participants
Groups:
- Adalimumab in Obese Participants: Obese participants were defined as having a BMI ≥ 30. Adalimumab was administered as follows: 80 mg at baseline, followed by 40 mg every other week (eow; starting at Week 1 until Week 15). The study drug was self-administered via subcutaneous (sc) injection.
- Adalimumab in Non-obese Participants: Non-obese participants were defined as having a BMI < 30. Adalimumab was administered as follows: 80 mg at baseline, followed by 40 mg every other week (eow; starting at Week 1 until Week 15). The study drug was self-administered via subcutaneous (sc) injection.
Arm/Group | Adalimumab in Obese Participants | Adalimumab in Non-obese Participants
Number analyzed (Participants) | 66 | 84
percentage of participants
  PASI-75 | 76 | 92
  DLQI <6 | 80 | 90

16. Secondary Outcome: Percentage of Obese vs. Non-obese (Per Waist-Hip Ratio) Participants Achieving a Psoriasis Area and Severity Index (PASI)-75 Response and a Total Dermatology Life Quality Index (DLQI) Score of <6 at Week 16
Description: The Waist-Hip Ratio was used to determine the groups of participants who were overweight and who were considered obese. Obesity was defined as a ratio of >1 for men and >0.8 for women. Response to treatment in participants with obesity (based on Waist-Hip Ratio) versus those without obesity was assessed via PASI-75 response (see Outcome Measure 1 for details) and DLQI score of <6 (see Outcome Measure 3 for details).
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Groups:
- Adalimumab in Obese Participants: Obese participants were defined as those with a waist-hip ratio of >1 for men and >0.8 for women. Adalimumab was administered as follows: 80 mg at baseline, followed by 40 mg every other week (eow; starting at Week 1 until Week 15). The study drug was self-administered via subcutaneous (sc) injection.
- Adalimumab in Non-obese Participants: Non-obese participants were defined as those with a waist-hip ratio of ≤1 for men and ≤0.8 for women. Adalimumab was administered as follows: 80 mg at baseline, followed by 40 mg every other week (eow; starting at Week 1 until Week 15). The study drug was self-administered via subcutaneous (sc) injection.
Arm/Group | Adalimumab in Obese Participants | Adalimumab in Non-obese Participants
Number analyzed (Participants) | 66 | 84
percentage of participants
  PASI-75 | 77 | 91
  DLQI <6 | 84 | 87

17. Secondary Outcome: Serum Levels of Folic Acid at Baseline and Week 4
Description: Normal values for folic acid were 3-15 ng/mL.
Time Frame: Baseline, Week 4
Population: Participants with available data at given time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Adalimumab
Number analyzed (Participants) | 143
ng/mL
  Baseline | 18.1 (20.0)
  Week 4 | 17.8 (11.4)

18. Secondary Outcome: Serum Levels of Vitamin B6 at Baseline and Week 4
Description: Normal values for vitamin B6 were 18-175 nmol/L.
Time Frame: Baseline, Week 4
Population: Participants with available data at given time points.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 141
nmol/L
  Baseline | 11.2 (12.5)
  Week 4 | 11.7 (11.6)

19. Secondary Outcome: Serum Levels of Vitamin B12 at Baseline and Week 4
Description: Normal values for vitamin B12 were 200-1100 pg/mL.
Time Frame: Baseline, Week 4
Population: Participants with available data at given time points.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Adalimumab
Number analyzed (Participants) | 143
pg/mL
  Baseline | 542.6 (615.5)
  Week 4 | 439.6 (438.9)

20. Secondary Outcome: Serum Levels of Folic Acid at Baseline and Week 16
Description: Normal values for folic acid were 3-15 ng/mL.
Time Frame: Baseline, Week 16
Population: Participants with available data at given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Adalimumab
Number analyzed (Participants) | 140
ng/mL
  Baseline | 18.2 (20.2)
  Week 16 | 17.9 (7.1)

21. Secondary Outcome: Serum Levels of Vitamin B6 at Baseline and Week 16
Description: Normal values for vitamin B6 were 18-175 nmol/L.
Time Frame: Baseline, Week 16
Population: Participants with available data at given time points.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 138
nmol/L
  Baseline | 11.4 (12.6)
  Week 16 | 11.8 (7.6)

22. Secondary Outcome: Serum Levels of Vitamin B12 at Baseline and Week 16
Description: Normal values for vitamin B12 were 200-1100 pg/mL.
Time Frame: Baseline, Week 16
Population: Participants with available data at given time points.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Adalimumab
Number analyzed (Participants) | 140
pg/mL
  Baseline | 541.9 (620.5)
  Week 16 | 441.8 (533.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of study through 70 days after the last treatment. Treatment duration was 15 weeks.
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 1/150
Other Adverse Events (participants affected / at risk) | 86/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=150)
Cholelithiasis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=150)
Anemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 1
Polycythemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Aortic arteriosclerosis (Cardiac disorders) | 1
Chest pain precordial (Cardiac disorders) | 1
Hypertension aggravated (Cardiac disorders) | 1
Otitis externa (Ear and labyrinth disorders) | 1
Otitis media (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Corneal injury (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Cholelithiasis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Epigastric discomfort (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Food poisoning (Gastrointestinal disorders) | 1
Gastrointestinal infection (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Oral infection (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Calculus urethral (Renal and urinary disorders) | 1
Nefrolithiasis (Renal and urinary disorders) | 1
Penis disorder (Renal and urinary disorders) | 1
Prostatitis (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Vaginal infection (Infections and infestations) | 1
C-Reactive Protein increase (Metabolism and nutrition disorders) | 2
Diabetes (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 16
Hypertransaminasemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 7
Hypervitaminosis B12 (Metabolism and nutrition disorders) | 3
Hypervitaminosis B6 (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2
Weight loss (Metabolism and nutrition disorders) | 1
Ankle sprain (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint injury (Musculoskeletal and connective tissue disorders) | 1
Anxiety (Psychiatric disorders) | 1
Seizures (Nervous system disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 8
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 6
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 17
Cold sores (herpetic) (Skin and subcutaneous tissue disorders) | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Papillomatosis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Application site pain and/or pruritus (General disorders) | 7
Fatigue (General disorders) | 4
Fever (General disorders) | 1
Pruritus generalized (General disorders) | 1
Psoriasis aggravated (General disorders) | 2
Skin disorder (General disorders) | 1
Skin nodule (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.